CLINICAL TRIAL: NCT05589116
Title: Investigating the Efficacy of a Two-week, Online Compassionate Imagery Intervention for Improving Mental Wellbeing in Veterinarians: A Randomised Controlled Trial
Brief Title: An Online Compassionate Imagery Intervention for Veterinarian Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FHMS 21022 252 EGA
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Compassion; Perfectionism; Rumination; Self-Criticism; Resilience
MeSH Terms: conditions — Rumination Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either a treatment or wait-list control group. The study will use a repeated measures, randomised controlled trial design.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants given immediate access to two-week, online compassionate imagery course.
  Interventions: Other: Online Compassionate Imagery Intervention
- Wait-list control group (No Intervention): Participants will not access intervention during 10-week study period (access will be given to online compassionate imagery course after all outcome measures have been completed).

INTERVENTIONS:
Other: Online Compassionate Imagery Intervention — The intervention comprises 14 pre-recorded, 10-15 minute videos. Participants will be asked to watch one video per day over a two-week period. The videos initially focus on providing psychoeducation about what self-compassion is, before delivering a series of guided Compassion Focused Therapy (CFT) informed exercises to cultivate self-compassion. The first week of the intervention will teach key compassion skills, with the second week focusing on skill consolidation.
  Arms: Intervention group

SUMMARY:
This randomised control trial aims to determine the efficacy of a two-week, online compassionate imagery intervention on improving veterinarian mental wellbeing. Participants will be randomly allocated to receive the intervention immediately or after a 10-week study period. Self-report questionnaires will be used at four time points to measure change on a range of psychological variables.

DETAILED DESCRIPTION:
Background: Research suggests that veterinarians are high-achievers with self-critical, perfectionist tendencies (Holden, 2020). Perfectionism in veterinarians has been associated with stress, anxiety, negative affect and low resilience (Crane, Phillips & Karin, 2015). However, McArthur et al. (2017) found that veterinarians with higher levels of self-compassion reported greater resilience. A feasibility study by Wakelin, Perman and Simonds (2022) found an online two-week compassion-focused imagery intervention to be acceptible and feasible for a veterinarian sample. Wakelin et al. (2022) also reported indications of preliminary effect as veterinarians illustrated a reduction in perfectionism, work-related rumination and self-criticism over the intervention period.

Aim: This study aims to extend Wakelin et al.'s (2022) research, to determine the efficacy of a two-week, online compassionate imagery intervention on improving veterinarian mental wellbeing.

Design: The study will use a mixed-methods, repeated measures, randomised controlled trial design.

The independent variables will be the intervention group (either treatment or wait list control) and the data collection time point. Six questionnaires will be used to collect quantitative data on the following dependent variables: perfectionism, work- related rumination, fear of compassion, resilience, self-compassion, self- criticism and self-reassurance.

Method: Participants will complete questionnaire measures at four time points: prior to randomisation (baseline), two weeks post-randomisation (post-intervention), six-weeks post-randomisation (one-month intervention follow-up) and ten-weeks after randomisation (two-month intervention follow up). Participants in the treatment group will be asked to watch a 10-15 minute compassionate imagery video every day for two weeks (14 in total). Participants in the control group will gain access to intervention materials upon study completion but their engagement in the videos will not be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Any student, recent graduate or qualified veterinary surgeon will be eligible for participation in the study.

Exclusion Criteria:

* Veterinarians who participated in Wakelin et al.'s (2022) feasibility trial.
* Veterinarians who are currently receiving a compassion- or cognitive-based therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Change in 'Functions of Self-Criticising/Attacking and Self-Reassuring Scale' (FSCRS; Gilbert, Clarke, Hempel, Miles & Irons, 2004). | 4 time points: baseline, immediate post-intervention, four weeks post-intervention and eight weeks post-intervention
  This 22-item scale will be used to measure self-criticism and self-reassurance. Participants are required to respond to statements on a 5-point Likert scale, ranging from 0 ('not at all like me') - 4 ('extremely like me'). The FSCRS has 3 subscales (Hated Self, Inadequate Self and Reassured Self) which are used to produce an overall self-criticism score (calculated by summing the Hated Self and Inadequate Self items) and a self-reassurance score (calculated by summing the Reassured Self items).

SECONDARY OUTCOMES:
Change in 'Brief Resilience Scale' (BRS; Smith et al., 2008) | 4 time points: baseline, immediate post-intervention, four weeks post-intervention and eight weeks post-intervention
  This 6-item scale will be used to measure resilience. The scale uses a combination of positively and negatively worded statements, which participants must respond to on a Likert Scale ranging from 1 ('strongly disagree') to 5 ('strongly agree'). The scores are summed to produce a total score, with a higher total score reflecting a higher level of resilience.
Change in 'Compassionate Engagement and Action Scales' Self-Compassion scale (CEAS; Gilbert et al., 2017) | 4 time points: baseline, immediate post-intervention, four weeks post-intervention and eight weeks post-intervention
  The 13-item CEAS Self-Compassion scale will be used to measure self-compassion. It uses a series of statements, to which the participant must respond on a Likert Scale with responses ranging from 1 ('never') to 10 ('always'). The scale has two subscales, which are aligned with the two dimensions of Gilbert's (2017) model of compassion: 'Compassionate Engagement' and 'Compassionate Action'. A total score can be produced by summing the subscale scores, with a higher score reflecting a higher level of self-compassion.
Change in 'Work-related Rumination Questionnaire' (WRRQ; Cropley, Michalianou, Pravettoni & Millward, 2012) | 4 time points: baseline, immediate post-intervention, four weeks post-intervention and eight weeks post-intervention
  This 25-item scale will be used to measure a person's tendency to engage in ruminative thinking about work; participants will be asked to respond in relation to their university, placement, or clinic work. The WRRQ has three subscales (affective rumination, problem-solving pondering, and distraction detachment), and a mean total score is calculated, with higher scores indicating a higher level of rumination.
Change in 'Frost Multidimensional Perfectionism Scale - 24 Items' (FMPS-24; Khawaja & Armstrong, 2005). | 4 time points: baseline, immediate post-intervention, four weeks post-intervention and eight weeks post-intervention
  This 24-item scale will be used to measure perfectionism. The scale is scored out of 120, with a higher score indicating stronger perfectionistic tendencies.
Change in 'Fears of Compassion Scale' (FCS; Gilbert, McEwan, Matos & Rivis, 2011). | 4 time points: baseline, immediate post-intervention, four weeks post-intervention and eight weeks post-intervention
  This 38-item scale will be used to measure Fears of Compassion and it comprises three subscales: Fears of Compassion-Self, Fears of Compassion- For others, and Fears of Compassion- From others.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Surrey, Guildford, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wakelin KE, Perman G, Simonds LM. Feasibility and efficacy of an online compassion-focused imagery intervention for veterinarian self-reassurance, self-criticism and perfectionism. Vet Rec. 2023 Jan;192(2):e2177. doi: 10.1002/vetr.2177. Epub 2022 Sep 10. PMID 36087064
- [Background] Holden CL. Characteristics of Veterinary Students: Perfectionism, Personality Factors, and Resilience. J Vet Med Educ. 2020 Jul;47(4):488-496. doi: 10.3138/jvme.0918-111r. Epub 2020 May 15. PMID 32412364
- [Background] Crane MF, Phillips JK, Karin E. Trait perfectionism strengthens the negative effects of moral stressors occurring in veterinary practice. Aust Vet J. 2015 Oct;93(10):354-60. doi: 10.1111/avj.12366. PMID 26412116
- [Background] McArthur M, Mansfield C, Matthew S, Zaki S, Brand C, Andrews J, Hazel S. Resilience in Veterinary Students and the Predictive Role of Mindfulness and Self-Compassion. J Vet Med Educ. 2017 Spring;44(1):106-115. doi: 10.3138/jvme.0116-027R1. PMID 28206835